CLINICAL TRIAL: NCT02514811
Title: Northwest Coalition for Adolescent Health (NWCAH) Teen Outreach Program Replication Study
Brief Title: Replication of the Teen Outreach Program in the Pacific Northwest
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philliber Research & Evaluation (Other)
Collaborators: Northwest Coalition of Adolescent Health (Unknown); The Office of Adolescent Health, HHS (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Philliber10-15ppgnw
Record Dates: First submitted 2015-07-27; First posted 2015-08-04 (Estimated); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Teenage Pregnancy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- The Teen Outreach Program (Experimental): TOP is a youth development and service learning program for youth designed to reduce teenage pregnancy and increase school success by helping youth develop a positive self-image, life management skills, and realistic goals. The TOP program model consists of three components implemented in school, after school, or in community settings over nine months: (1) weekly curriculum sessions, (2) community service learning, and (3) positive adult guidance and support. The TOP Changing Scenes Curriculum is separated into four age-/stage-appropriate levels, Level 1 is typically for youth ages 12 or 13 and Level 4 is typically for youth age 17. The intended program dosage for each participant is a minimum of 25 weekly sessions and at least 20 hours of community service learning over nine months. One or two facilitators, who plan the order of sessions based on the needs and interest of youth, implemented TOP in a group of 10 to 25 youth.
  Interventions: Behavioral: The Teen Outreach Program
- Control Group (No Intervention): Students in the control condition receive a benign intervention called the Community Voices (CV) program, which like TOP, meets in a group setting. The CV students are convened four times during the program year. Sessions are the same length as the TOP sessions. The first and last CV sessions are primarily focused on survey data gathering. At the two other sessions, CV students are convened to discuss current issues among young people in their community. The CV program specifically does not include any sexuality education or community service learning opportunities.

INTERVENTIONS:
Behavioral: The Teen Outreach Program — Students received the Teen Outreach Program as described previously.
  Arms: The Teen Outreach Program

SUMMARY:
The Northwest Coalition for Adolescent Health (NWCAH) replicated the Teen Outreach Program (TOP) in five states across the pacific northwest including Idaho, Alaska, Montana, Oregon, and Washington. The purpose of this study is to measure: at the end of the program year, were TOP students less likely than control group students to report ever being pregnant or causing someone to be pregnant?

ELIGIBILITY:
Inclusion Criteria:

* Has parental consent and student assent
* Attends one of the schools and/or classes chosen for the program

Exclusion Criteria:

* Lack of consent or assent

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 8686 (Actual)
Dates: Start 2011-09; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
Pregnancies | 9 months
  In the spring at the end of the program year, did the Teen Outreach Program students report significantly fewer pregnancies or births than the students in the Community Voices (the counterfactual) program?

SECONDARY OUTCOMES:
Pregnancies at follow up | 21 months
  In the spring, one year following the end of the program year, did the Teen Outreach Program students report significantly fewer pregnancies or births than the students in the Community Voices (the counterfactual) program?
Sexual behavior | 9 months
  In the Spring, at the end of the program year, what is the impact of the Teen Outreach program relative to the Community Voices program (the counterfactual) on sexual behavior?
Contraceptive use | 9 months
  In the Spring, at the end of the program year, what is the impact of the Teen Outreach program relative to the Community Voices program (the counterfactual) on contraception use?

CONTACTS AND LOCATIONS:
Overall Officials: Susan Philliber, PhD, Principal Investigator — Philliber Research Associates